CLINICAL TRIAL: NCT04467242
Title: Interaction Between Right Heart Dysfunction and Emphysema: Impact of Endoscopic Lung Volume Reduction (RVDD)
Brief Title: Right Ventricular Diastolic Dysfunction
Acronym: RVDD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0372
Record Dates: First submitted 2020-07-01; First posted 2020-07-10 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-06

CONDITIONS: COPD; Emphysema; Right Heart Dysfunction
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COPD patients: COPD patients with severe emphysema and right heart dysfunction

SUMMARY:
Heart-lung interactions remain misunderstood whereas pulmonary and cardiac pathologies are very commonly associated.

Emphysema by increasing intrathoracic pressure appears to affect cardiac function.

Interestingly, previous studies have shown a link between the telediastolic volume of the right ventricle (measured by RMI) and the intensity of emphysema.

Our hypothesis is that the emphysema by increasing intrathoracic pressure leads to or accentuates right cardiac diastolic dysfunction by decreasing compliance and cardiac preload.

To verify this hypothesis the investigators will perform KT loop procedures in order to acquire intracardiac pressure/volume curves before and after lung volume reduction.

The pressure/volume curves allow the analysis of systolic and diastolic function, cardiac contractility and loading conditions.

ELIGIBILITY:
Inclusion criteria:

* At least 40 years
* A smoking history
* Smoking cessation ≥ 6 months
* FEV1/FVC ≤ 0,7
* Severe emphysema (destruction ≥ 50%)
* Peak tricuspid regurgitation velocity < 2,8 m/s or presence of other echocardiographic "PH signs"
* 15% ≤ FEV1post ≤ 50%
* Residual volume ≥ 175% predicted
* TLC ≥ 100% predicted
* Optimal medical management
* 150m ≤ 6MWD ≤ 500m
* mMRC ≥ 2
* Physical activity ≥ 2/Week (≥ 30minutes)

Exclusion criteria:

* ≥2 hospitalizations/year for EACOPD
* Recent EACOPD (≤ 3months)
* ≥ 50ml mucus/day
* PAPm ≥35mmHg
* PaCO2 ≥ 55mmHg
* Bubble ≥ 1/3 hemithorax
* Lung fibrosis, bronchiectasis, lung cancer, homolateral surgery
* Left ventricular ejection fraction ≤ 45%, unstable heart disease
* Life expectancy ≤ 1 year
* Contraindication to anesthesia
* Allergy to nitinol or silicone
* Corticotherapy ≥ 10mg/day
* Patient under legal protection

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients with severe emphysema and right heart dysfunction
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-07-20 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Estimate the change in right diastolic cardiac function after reduction of emphysema | 1 day
  Estimate the change in right diastolic cardiac function after reduction of emphysema : assessed by the change in the slope end diastolic pressure volume relationship (EDPVR mmHg/ml) obtained by KT Loop procedure

SECONDARY OUTCOMES:
Estimate the change in right systolic heart function | 1 day
  Estimate the change in right systolic heart function before and after reduction of emphysema assessed by the cardiac output (L/min), the stroke volume (ml), the end systolic pressure (mmHg), the end systolic volume (mmHg), obtained by KT Loop procedure
Estimate the change in right cardiac contractility | 1 day
  Estimate the change in right cardiac contractility before and after reduction of emphysema assessed by the slope end systolic pressure volume relationship (mmHg/ml), obtained by KT Loop procedure.
Estimate ventriculo-arterial coupling | 1 day
  Estimate ventriculo-arterial coupling before and after reduction of emphysema assessed by the Ees/Ea ratio, obtained by KT Loop procedure
Evaluate the evolution of symptoms assessed | 1 day
  Evaluate the evolution of symptoms assessed by the Mmrc questionnaire and the CATCOPD questionnaire before and after reduction of emphysema.
Assessing exercice performance | 1 day
  Assessing exercice performance by the 6 minutes walk test before and after reduction of emphysema.
Evaluate the evolution of respiratory function | 1 day
  Evaluate the evolution of respiratory function before and after reduction of emphysema assessed by the FEV1 (Liters and % of predicted value), the FVC (Liters and % of predicted value), the RV (Liters and % of predicted value), the TLC (Liters and % of predicted value) obtained by spirometry/plethysmography.

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Bourdin, MD PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC